CLINICAL TRIAL: NCT02950649
Title: Evaluation of Clinical Impact of Non-Invasive Hemodynamic Monitoring to Optimize Perioperative Care in Moderate to High Risk Patients With Poor Functional Status
Brief Title: Evaluation of Clinical Impact of Non-Invasive Hemodynamic Monitoring to Optimize Perioperative Care
Status: Terminated | Type: Observational
Why Stopped: PI left institution 10/01/2020 and no further subjects were enrolled and no further data was collected.
Sponsor: Loma Linda University (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Melissa McCabe, Assistant Professor Cardiothoracic Anesthesiology, Loma Linda University
Other Study IDs: 5160227
Record Dates: First submitted 2016-08-03; First posted 2016-11-01 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Hemodynamic Monitored Guided Assesment: This group will have the non-invasive hemodynamic monitoring device placed and the data will be used for comparison with routine subjective preoperative assessment assessment.
  Interventions: Device: invasive Hemodynamic monitoring via Clearsight/Nexfin Systems from Edwards Lifesciences
- No Hemodynamic Monitored Guided Assesment: This group will have subjective assessment by the provider and this data will be compared to the device assessment of cardiac index..
  Interventions: Device: No Hemodynamic Monitored Guided Assesment

INTERVENTIONS:
Device: invasive Hemodynamic monitoring via Clearsight/Nexfin Systems from Edwards Lifesciences — Experimental: Hemodynamic Monitored Guided Assesment This group will have the non-invasive hemodynamic monitoring device placed and its data will help guide (intervention) patient's management decisions (experimental).
  Groups: Hemodynamic Monitored Guided Assesment
Device: No Hemodynamic Monitored Guided Assesment — Arm: Active Comparator: No Hemodynamic Monitored Guided Assesment This group will have the non-invasive hemodynamic monitoring device placed but its data will NOT be factored for intervention of the patient's management decisions.
  Groups: No Hemodynamic Monitored Guided Assesment

SUMMARY:
This project is designed to assess the impact of pre-operative use of non-invasive hemodynamic monitoring technologies on improving peri-operative and post-operative care of moderate to high-risk surgical patients with poor functional status by improving the detection of reduced cardiovascular function.

DETAILED DESCRIPTION:
This study seeks to evaluate the impact of using a non-invasive technology to assess flow guided parameters (SV,SVR, dp/dt, CO, etc.) on patient care decisions in the preoperative settings. Patients seen in the preoperative clinic who are undergoing a moderate or high-risk procedure and have less than 4 metabolic equivalents (METs) will be approached to participate in the study .

Once consented, the device will be placed during the preoperative clinic visit and the data will be presented to the care team. Surveys will be completed by the health care provider for each consented patient to determine if the data from the device positively impacted patient care decisions. Specifically, the survey will evaluate if providing information on the patient's cardiovascular function (via the device used for this study) facilitated the health care provider to identify if the patient had reduced cardiovascular function. For the primary outcome, this study will evaluate if this device can assistant the identification of patients with reduced cardiovascular function by providing the flow guided parameter listed above. Secondary markers include the evaluation of perioperative complication rate (composite outcome ) between those that had the non-invasive HD data displayed to the preoperative team vs. not. Additional secondary makers will include: frequency of intraoperative hemodynamic optimization and goal directed fluid therapy administration, health care provider survey results, patient survey on the level of discomfort from wearing the cuff during the study. length of hospital stay, length of intensive care stay, readmission to the hospital within 30 days after hospital discharge, and 30-day postoperative mortality.

Outcome data will be collected using the electronic medical records database available at the investigators institution.

It is the hope of the investigators that this study will demonstrate that by simply applying the preoperative use of the non-invasive hemodynamic technologies one can:

1. more appropriately identify which patients would benefit from intraoperative hemodynamic monitoring strategies
2. increase satisfaction of the preoperative assessment by the health care provider
3. further validate the importance of caring for patients with knowledge of their volume status, contractility, and vascular resistance in other patient care settings.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (greater than 18 years of age)
2. ASA classification 3 and 4 level patients with poor functional status,
3. less than 5 metabolic equivalents (METs) -

Exclusion Criteria:

1. < 18 years of age, pregnancy,
2. known severe peripheral artery disease,
3. poor perfusion to fingers (as defined as a perfusion index less than 0.5%- www.Masimo.com),
4. history of Raynaud's,
5. refusal to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with ASA classification level 3 and 4, with less than 5 metabolic events
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of subjective assessment compared to device assessment of cardiac index | Up to one year from date of randomization
  Comparison of cardiac index derived from subjective preoeprative assessment to cardiac index derived from device assessment

CONTACTS AND LOCATIONS:
Overall Officials: Davinder Ramsingh, MD, Principal Investigator — Loma Linda University Health
Locations (3):
- United States (3):
  - Loma Linda Health, Loma Linda, California
  - Loma Linda University Department of Anesthesiology, Loma Linda, California
  - Pat Moore, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No